CLINICAL TRIAL: NCT00206791
Title: Study of Osteoconduction Potential of an Injectable Calcium Phosphate in Orthopaedic Surgery in Fillings of Osseous Defects From Various Origins
Brief Title: Osteoconduction Potential of an Injectable Calcium Phosphate in Orthopaedic Surgery in Fillings of Osseous Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomatlante (Industry)
Responsible Party: Pr CATONNE, CHU Bordeaux
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002/01/001
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2006-10

CONDITIONS: Grafting, Bone
Keywords: bone substitutes; Bone Replacement Materials; bone void filler; Grafting, Bone; Bone Cysts
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBCPGel (Experimental)
  Interventions: Device: MBCP-Gel (tm); Device: MBCP Gel

INTERVENTIONS:
Device: MBCP-Gel (tm) — MBCPGel 5ml
  Other Names: injectable resorbable biphasic calcium phosphate
Device: MBCP Gel — MBCPGel 5ML
  Other Names: Injectable biphasic calium phosphate

SUMMARY:
The purpose of this non-comparative study is to test, for the first time, the bioactivity of a new "ready to use" calcium phosphate biomaterial in fillings of little losses of osseous substance from various origins, such as traumatic and benign tumoral causes.

DETAILED DESCRIPTION:
A lot of osseous substitution products were already used to fill osseous defects in order to prevent losses of osseous that are envisaged and so prejudicial.

Synthetic calcium phosphate ceramics (particularly granulated forms) already has shown their osteoconduction potential in human at different sites. But it is difficult to put these granules in very little place.

The injectable form of calcium phosphate granules "ready to use" is easier to be used and allow a diminution of the risk of infection during surgery, and permit homogeneity of the biomaterial.

Injectable form of calcium phosphate granules did already has shown his biocompatibility and biofunctionality in animals.

The purpose of this study is to study the biocompatibility and biofunctionality of this biomaterial in his injectable form in fillings of little losses of osseous substance from various origins were no charge will act to the biomaterial.

ELIGIBILITY:
Inclusion Criteria:

* Medium osseous defects (inferior to 20 cc) without articular communication
* Patients without a personal medical history of bone infection, cancer, diabetes, tuberculosis, and in general, any pathology which could interfere with the results of the study or expose the patient to additional risk
* Patients without drepanocytosis, or congenital or acquired immunizing deficit
* Patients who have the benefit of a social security system, a previous medical exam and who were informed and gave free consent about this study

Exclusion Criteria:

* Proven nicotinism and alcoholism
* Pregnant or nursing women
* Patients who received another study drug or another study device in the past 3 months or patients who will be included in another clinical study
* If postoperative follow-up for a patient is considered to be random by the investigator, he/she should not be included

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Presence or absence of an edging to radiolucent on the radiographic stereotypes between the biomaterial and the osseous walls of the osseous defect at different times (3, 6 and 12 months after surgery) | 3, 6 and 12 months

SECONDARY OUTCOMES:
An analysis of numeric radiographic stereotypes by grey steps will study the evolution of the density of the implant and environmental bone. | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: CATONNE Y, Pr., Principal Investigator — Hôpital de la Pitié Salpétrière - 75013 PARIS - France
Locations (4):
- France (4):
  - CHU de Bordeaux - Hôpital PELLEGRIN -Service d'Orthopédie - Traumatologie C, Bordeaux
  - CH des Broussailes - Service de Chirurgie Orthopédique et Traumatologique, Cannes
  - CHU de Fort de France - Hôpital Pierre ZODBA-QUITMAN - Service d'Orthopédie et Traumatologie, Fort de France
  - Service de Chirurgie Orthopédique et Traumatologique - CHU de la Pitié Salpétrière, Paris